CLINICAL TRIAL: NCT00763100
Title: The Efficacy of Tomosynthesis in the BIRADS 3 Population Including Surveillance of Patients in the Treatment or Post-Treatment for Breast Cancer
Brief Title: Efficacy of Tomosynthesis in the BIRADS 3 Population
Acronym: BIRADS
Status: Completed | Type: Observational
Sponsor: WellSpan Health (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Joanne Trapeni, DO, Women's Imaging Center
Other Study IDs: 0708023
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Three dimensional versus two dimensional; Breast cancer surveillance; Tomosynthesis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Breast cancer: Patients in treatment or post-treatment for breast cancer

SUMMARY:
There are three main objectives, centering on those patients targeted for surveillance imaging. The first objective is to compare image quality and specificity of breast tomosynthesis and conventional 2D mammography in a BIRADS 3 diagnostic population. The second objective is to compare image quality and ability to determine post-surgical and post-radiation changes from recurrence in a post-cancer subset of a BIRADS 3 population having undergone conservation therapy (lumpectomy with or without radiation. The final objective is to compare image quality and the ability to determine chemoresponsiveness in a post-cancer subset of a BIRADS 3 population, who are undergoing neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

GROUP 1

* female of any race and ethnicity
* 35 years or older
* after routine and diagnostic imaging, subject is categorized as a BI-RADS 3 and will undergo study imaging within 30 days of routine or diagnostic imaging.
* subject is returning for surveillance imaging after a categorization of a BI-RADS 3 and will undergo study imaging within 30 days of surveillance imaging GROUP 2
* female of any race and ethnicity
* 26 years or older
* subject has completed cancer treatment and is currently categorized as a BI-RADS 3 for surveillance imaging
* subject will undergo study imaging within 30 days of surveillance imaging GROUP 3
* female of any race and ethnicity
* 26 years or older
* subject is currently undergoing cancer treatment and is currently categorized as a BI-RADS 3 for surveillance imaging OR
* subject will undergo study imaging within 30 days of surveillance imaging

Exclusion Criteria:

* GROUP 1, 2 and 3
* subjects unable or unwilling to participate
* subjects who are unable or unwilling to tolerate compression
* subjects who are pregnant or who think they may be pregnant
* subjects who are breastfeeding

Min Age: 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three groups of patients will be enrolled:
  Group 1 will enroll patients that have been categorized as a BIRADS 3 on the basis of screening and diagnostic conventional imaging work-up.
  Group II will enroll patients that have been categorized as a BIRADS 3 for surveillance imaging because they have undergone breast conservation therapy for breast cancer.
  Group III will enroll patients that have been categorized as a BIRADS 3 for surveillance imaging because they are currently undergoing primary systemic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 690 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
to see if Breast Tomosynthesis, a three-dimensional (3D) imaging study is more accurate than standard mammography (a two-dimensional (2D) study). | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Trapeni, DO, Principal Investigator — WellSpan Health